CLINICAL TRIAL: NCT06668714
Title: Does Co-administration of Lactate Affect Postprandial Nutrient Absorption and Fat Disposition?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Natasa Brkovic Zubanovic, Principal Investigator, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LAMETA-PET
Record Dates: First submitted 2024-09-17; First posted 2024-10-31 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pre Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Glucose Intolerance; Metabolic Syndrome | interventions — Lactic Acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo pre-diabetes (Placebo Comparator)
  Interventions: Combination Product: Placebo + mixed meal; Combination Product: Lactate + mixed meal; Radiation: PET-scan
- Lactate pre-diabetes (Experimental)
  Interventions: Combination Product: Placebo + mixed meal; Combination Product: Lactate + mixed meal; Radiation: PET-scan
- Healthy (Active Comparator): We will include 8 healthy, normal-weight individuals (BMI 20-25 kg/m2, age 50+ years) as a healthy control group, who will be studied twice following ingestion of a liquid test meal to determine the differences in meal fat partitioning between insulin-sensitive and insulin-resistant individuals and to determine the intraindividual variation in meal fat partitioning. Furthermore, the extra PET scans performed in the healthy individuals will be used for precise quantification of the radiation exposure with the PET method (dosimetry) and validation of the PET method.
  Interventions: Radiation: PET-scan; Combination Product: Mixed meal with 18F-FTHA

INTERVENTIONS:
Combination Product: Placebo + mixed meal — Placebo (140 mL isoosmotic salt water, NaCl) given 30 minutes before a liquid test meal with the addition of 70 MBq 18F-FTHA = CTR
  Arms: Lactate pre-diabetes; Placebo pre-diabetes
Combination Product: Lactate + mixed meal — Lactate (140 mL lactate drink = 25 g D/L-lactate bound to Na) given 30 minutes before a liquid test meal with the addition of 70 MBq 18F-FTHA = LAC The investigators will also use the 18F-FTHA standardized uptake value (SUV) to evaluate dietary fatty acid trapping and distribution, to be able to compare our results with former studies using the 18F-FTHA method.
  Arms: Lactate pre-diabetes; Placebo pre-diabetes
Radiation: PET-scan — Dynamic whole-body PET scan.
Combination Product: Mixed meal with 18F-FTHA — Mixed meal test with the addition of 70 MBq 18F-FTHA
  Arms: Healthy

SUMMARY:
Aim To investigate the effects of oral lactate administration on nutrient absorption and substrate utilization in individuals with pre-diabetes.

Hypothesis The addition of lactate to a meal improves postprandial lipemia and reduces lipid storage in ectopic tissues through delayed absorption and faster removal of circulating lipids from circulation.

DETAILED DESCRIPTION:
A recent study showed that oral lactate administration slowed gastric emptying, increased the feeling of being full, induced satiety, and decreased the anticipated future food intake compared with intravenous administration. This shows that lactate has direct effects in the GI tract, which could improve substrate utilization after meals and thereby improve metabolic health. However, it remains unknown whether oral lactate administration has similar effects in other populations (i.e. individuals with obesity) and in relation to a meal.

To address these potential effects, the investigators aim to implement and validate a new tracer method in Denmark to measure meal fat partitioning using an orally ingested fluorine-labeled fatty acid analog (18F-fluoro-6-thiaheptadecanoic acid, 18F-FTHA) combined with positron emission tomography coupled to computed tomography (PET-CT). In a previous study using the aforementioned method, it has been shown that individuals with an impaired glucose tolerance have increased myocardial fatty acid uptake, not explained by potential confounding factors and that this is associated with a reduced systolic ejection fraction. In a recent study, it was found that subjects with insulin resistance have a higher uptake of free fatty acids in visceral adipose tissue compared with subjects without insulin resistance.

This method will enable the investigators to determine how the addition of lactate to a test meal will affect meal fat partitioning. Previous methods for determining fatty acid partitioning and accumulation have either been limited to only determining the accumulation in non-oxidative tissues or very invasive or difficult to perform, making this the first method to non-invasively simultaneously measure the partitioning of meal fatty acids in all human organs.

Work package 1 (WP1):

The investigators will also include 8 healthy individuals (HbA1c mmol/mol< 39, age 50+ years) as a healthy control group, who will be studied twice in a randomized trial following ingestion of a liquid test meal to determine the differences in meal fat partitioning between insulin-sensitive and insulin-resistant individuals and to determine the intraindividual variation in meal fat partitioning. Furthermore, the extra PET scans performed in the healthy individuals will be used for precise quantification of the radiation exposure with the PET method (dosimetry) and validation of the PET method.

Work package 2 (WP2):

In a randomized, double-blinded placebo-controlled crossover trial, the investigators will investigate the effect of 25 g lactate vs. placebo prior to a liquid test meal, with the addition of 18F-FTHA, on two trial days separated by a minimum of seven days and a maximum of one month. The investigators will include 16 individuals with pre-diabetes (HbA1c 39-47 mmol/mol) and from 50+ years of age.

In a WP3 we will include one healthy participant who will receive 18F-FTHA with water instead of a mixed meal, to evaluate if the tracer can be used for diagnostics of lesions of the thoracic duct when given with water.

The investigators will use paired t-tests analyses for comparing CTR and LAC and independent t-test samples for comparing the individuals with pre-diabetes and the healthy individuals.

Based on the results from a previous study using 18F-FTHA-PET, the investigators will need to include 15 individuals to detect a 15% decrease in meal fat uptake in the heart (α=0.05, β=0.80). To account for potential missing values or failed PET-CT scans, the investigators will include a total of 16 individuals.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years
* Written and oral consent
* HbA1c 39-47 mmol/L

Exclusion Criteria:

* Medicine with an impact on blood glucose and glucose metabolism.
* Newly started medicine (<3 months prior to the inclusion time)
* Medicine changes (<3 months prior to the inclusion time and planned changes during the trial)
* Affected screening blood sample as evaluated by PI
* Hba1c > 47
* Allergy to paracetamol
* Doesn't speak or understand Danish
* Special diets

The eight healthy individuals will be included by the same criteria except for not having pre-diabetes

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Difference in meal fat uptake in heart tissue between CTR and LAC following a liquid test meal | 5-6 hours
  The investigators will use a dynamic whole-body PET scan to determine dietary fatty acid trapping and distribution by measuring available 18F-FTHA-tracer in blood coupled with measurement of radioactivity in different organs.
  The investigators will also use the 18F-FTHA standardized uptake value (SUV) to evaluate dietary fatty acid trapping and distribution, to be able to compare our results with former studies using the 18F-FTHA method.

SECONDARY OUTCOMES:
Difference in meal fat uptake in skeletal muscle, liver, subcutaneous fat, heart and visceral fat | 7 hours
  We will use a dynamic whole-body PET scan to determine dietary fatty acid trapping and distribution by measuring available 18F-FTHA-tracer in blood coupled with measurement of radioactivity in different organs.
  We will also use the 18F-FTHA standardized uptake value (SUV) to evaluate dietary fatty acid trapping and distribution, to be able to compare our results with former studies using the 18F-FTHA method.
Difference in absorption rate and distribution of free fatty acids. | 7 hours
  We will draw blood samples from arterialized blood from a perifery venous catheter and measure the concentration of free fatty acids on the two trial days.
Difference in subjective appetite sensation | 7 hours
  Subjective appetite sensation will be quantified using the appetite questionnaires consisting of a visual analog scale.
Difference in ventricular emptying rate | 7 hours
  We will use the acetaminophen test to evaluate ventricular emptying rate. The participants will drink 1500 mg paracetamol together with the mixed meal, and afterwards blood samples will be drawn and the concentration of acetaminophen will be measured during the trial day and compared between the two trial days.

CONTACTS AND LOCATIONS:
Overall Officials: Esben Søndergaard, Principal Investigator — Aarhus University, Steno Diabetes Center Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark